CLINICAL TRIAL: NCT00025766
Title: TOSCA-2: An Angiographic Substudy (Ancillary) of the Occluded Artery Trial (OAT)
Brief Title: Angioplasty and Heart Stents to Treat Individuals With an Occluded Artery Following a Heart Attack
Acronym: TOSCA-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Dr. Vladimir Dzavik, University Health Network, Toronto, ON, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 989; R01HL067683 (NIH)
Record Dates: First submitted 2001-10-22; First posted 2001-10-23 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction | interventions — Percutaneous Coronary Intervention; Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): PCI with stenting of the occluded culprit infarct-related artery plus optimal medical therapy
  Interventions: Device: PCI with stenting; Behavioral: Optimal Medical Therapy
- 2 (Active Comparator): Optimal medical therapy alone without PCI of the occluded culprit artery
  Interventions: Behavioral: Optimal Medical Therapy

INTERVENTIONS:
Device: PCI with stenting — PCI with stenting of the occluded culprit infarct-related artery
  Arms: 1
Behavioral: Optimal Medical Therapy — Participants will receive optimal medical therapy.

SUMMARY:
The purpose of this study is to evaluate arterial patency and left ventricular ejection fraction by examining angiographic data one year following a heart attack and treatment with late revascularization.

DETAILED DESCRIPTION:
BACKGROUND:

The Occluded Artery Trial (OAT) is an international study with 3200 participants. Its goal is to determine if delayed mechanical reperfusion by means of percutaneous transluminal coronary angioplasty (PTCA) and stenting reduces death, heart attacks, and hospitalization in individuals with New York Heart Association (NYHA) Class IV heart failure and a persistently occluded infarct-related artery (IRA) 3 to 28 days following a heart attack. While left ventricular (LV) function improvement has been suggested as a benefit of late reperfusion, solid evidence to support this claim is lacking. Furthermore, while stenting has reduced reocclusion rates after total occlusion PTCA, the reocclusion rate after a recent heart attack is unknown.

DESIGN NARRATIVE:

This study is a substudy of OAT and will enroll 380 participants. The primary aims of the study include the following: 1) to compare long-term patency rates between the two treatment groups (conventional medical therapy or PTCA and stenting) by means of follow-up coronary angiography one year after enrollment; and 2) to compare the change in global LV ejection fraction between the two treatment groups utilizing baseline and follow-up contrast LV angiograms. Secondary aims include the following: 1) comparison of regional wall motion and LV volumes; 2) study of the effect of reocclusion and spontaneous recanalization on LV function; and 3) study of the effect of duration of occlusion on changes in LV function after Percutaneous Coronary Intervention (PCI). The substudy will be conducted at 21 OAT study sites. The Substudy Coordinating Center (SCC) is at the University of Alberta in Edmonton, Canada. The Data Coordinating Center (DCC) is at the Maryland Medical Research Institute, which is the DCC for the OAT study. The Angiographic Core Laboratory is at the University of British Columbia.

ELIGIBILITY:
Inclusion Criteria:

* Has experienced a heart attack 3 to 28 days prior to study entry
* Has a persistently occluded IRA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2001-09; Primary Completion 2006-04 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
LV ejection fraction | 1 year
Infarct-related artery patency (measured by contrast LV and coronary angiography) | 1 year

SECONDARY OUTCOMES:
Comparison of regional wall motion and LV volumes | 1 year
Effect of reocclusion and spontaneous recanalization on LV function | 1 year
Effect of duration of occlusion on changes in LV function after PCI | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Dzavik, MD, Study Chair — University Health Network - Toronto General Hospital
Locations (1):
- University Health Network - Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Dzavik V, Buller CE, Lamas GA, Rankin JM, Mancini GB, Cantor WJ, Carere RJ, Ross JR, Atchison D, Forman S, Thomas B, Buszman P, Vozzi C, Glanz A, Cohen EA, Meciar P, Devlin G, Mascette A, Sopko G, Knatterud GL, Hochman JS; TOSCA-2 Investigators. Randomized trial of percutaneous coronary intervention for subacute infarct-related coronary artery occlusion to achieve long-term patency and improve ventricular function: the Total Occlusion Study of Canada (TOSCA)-2 trial. Circulation. 2006 Dec 5;114(23):2449-57. doi: 10.1161/CIRCULATIONAHA.106.669432. Epub 2006 Nov 14. PMID 17105848
- [Result] Steigen TK, Buller CE, Mancini GB, Jorapur V, Cantor WJ, Rankin JM, Thomas B, Webb JG, Kronsberg SS, Atchison DJ, Lamas GA, Hochman JS, Dzavik V. Myocardial perfusion grade after late infarct artery recanalization is associated with global and regional left ventricular function at one year: analysis from the Total Occlusion Study of Canada-2. Circ Cardiovasc Interv. 2010 Dec;3(6):549-55. doi: 10.1161/CIRCINTERVENTIONS.109.918722. Epub 2010 Nov 9. PMID 21062997
- [Result] Dzavik V, Buller CE, Devlin G, Carere RG, Mancini GB, Cantor WJ, Buszman PE, Rankin JM, Vozzi C, Ross JR, Forman S, Barton BA, Lamas AG, Hochman JS. Angiographic and clinical outcomes of drug-eluting versus bare metal stent deployment in the Occluded Artery Trial. Catheter Cardiovasc Interv. 2009 May 1;73(6):771-9. doi: 10.1002/ccd.21930. PMID 19309733